CLINICAL TRIAL: NCT00751010
Title: Relationship: Interstitial Cystitis & Vulvodynia-Part 2
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Donna Carrico, NP, William Beaumont Hospital
Other Study IDs: 2008-139
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Vulvodynia
Keywords: Vulvar pain; Vulvodynia; Interstitial cystitis
MeSH Terms: conditions — Vulvodynia; Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: In a mailed survey (Part 1 of this study), 127 women with a documented diagnosis of IC agreed to be contacted for an in-office examination.

SUMMARY:
The etiology of pain in women with IC is often difficult to identify resulting in unnecessary medical and surgical treatments (e.g. hysterectomies). The vulva may actually be the site of some of the reported pain in women with IC, not the urethra or bladder. IC and vulvodynia can impact one's sexual functioning and diminish one's quality of life. Unfortunately, vulvodynia is often unrecognized since it is not part of the usual urological assessment with IC patients.

Vulvodynia is characterized by persistent generalized or localized vulvar pain of varying degrees often characterized as "burning," suggestive of a neuropathic pain response.

DETAILED DESCRIPTION:
In a mailed survey (Part 1 of this study), 127 women with a documented diagnosis of IC agreed to be contacted for an in-office examination. The mailed survey was internally developed specifically for this project and included items related to demographics, adolescent and adult history related to genital pain and current health. The last section allowed the subject to include contact information if they would also like to participate in Part 2 (additional questionnaires and examination) of the study.

The study coordinator will review those surveys containing contact information and all women at least 18 years of age will be invited to the WISH program (Beaumont Women's Initiative for Pelvic Pain and Sexual Health) to be examined by a certified Nurse Practitioner (NP) who will be blinded to their survey responses.

Questionnaires will be completed by the subject. These questionnaires relate to one's history, pain symptoms, quality of life, bladder symptoms and sexual function and will be completed prior to the examination. The NP will perform all the clinical evaluations. A vaginal pH and wet mount slide will be done first. Testing for vulvodynia will be done utilizing an algesiometer q-tip followed by Neurometer® surface CPT testing for pain threshold (not tolerance) to quantify pain levels in the distribution of the pudendal nerve on the perineum and vulva will be done. The Neurometer® current perception threshold (CPT) is a device for evaluating and measuring sensation It is a battery-operated stimulator which delivers painless electrical stimulation via surface electrodes at frequencies of 5 Hz, 250 Hz, and 2000 Hz and at a current of 0.01 to 99mAmps.

ELIGIBILITY:
Inclusion Criteria

* Women with interstitial cystitis and vulvar pain who agreed to be contacted in Part 1 (HIC #2007-183) of this study.
* Age 18 or older
* Capable of giving informed consent
* Capable and willing to follow all study procedures

Exclusion Criteria:

* Pregnant women· Vaginitis (may be treated, then tested later)
* Vulvar disease (other than vulvodynia)-lichen planus, lichen sclerosis, neoplasia
* The subject is deemed unsuitable for enrollment by the investigators based on their history or physical examination.
* Neuropathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received a mailed survey (Part 1 of this study), with a documented diagnosis of IC who agreed to be contacted for an in-office examination.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The objective of our study is to identify and clinically confirm the presence of vulvodynia in women diagnosed with Interstitial Cystitis (IC) based on mailed survey results (Part 1, HIC #2007-183) and confirmed with a clinical assessment. | Visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Donna Carrico, NP, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States